CLINICAL TRIAL: NCT06209515
Title: Sociodemographic Factors and Criminal Behaviour Preceding Neurodegenerative Disease - Retrospective Register Study
Acronym: DEGERWD
Status: Active, not recruiting | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DEGERWD
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Neurodegenerative Diseases; Alzheimer Disease; Frontotemporal Dementia; Lewy Body Disease; Vascular Dementia; Parkinson Disease; Progressive Supranuclear Palsy; Corticobasal Degeneration; Multiple System Atrophy; Amyotrophic Lateral Sclerosis; Huntington Disease
MeSH Terms: conditions — Neurodegenerative Diseases; Alzheimer Disease; Frontotemporal Dementia; Lewy Body Disease; Dementia, Vascular; Parkinson Disease; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Multiple System Atrophy; Amyotrophic Lateral Sclerosis; Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with neurodegenerative disease: Patient diagnosed with neurodegenerative disease (ICD-10 diagnosis code) between 2010-2021
- Matched controls: Age, gender, and place of residency matched for those of a patient that was alive at the end of the year of the diagnosis

SUMMARY:
In this retrospective register study, clinically classified individuals with neurodegenerative disease from the years 2010-2021 will be verified from the clinical records from KUH and Oulu University Hospital (OUH). Based on the Finnish social security number, these individuals will be linked to the the national registers of Statistics Finland and Finnish Social and Health Data Permit Authority Findata including incomes, sociodemographic factors, education, occupation, criminal records as well as to the national registers including the bought pharmaceuticals, comorbidities and causes of death. For each study case, 10 randomly selected control cases, matched with age, sex and geographical area, will be used.

The aim of the study is to examine:

* 1) The prevalence of criminal and other disruptive behaviour in groups of different neurodegenerative diseases prior to and after the diagnosis
* 2) Changes in employment, residency,income, and marital status prior to and after the neurodegenerative disease diagnosis
* 3) Hospital diagnoses and reimbursable drugs prior to and after the diagnosis
* 4) Causes of death in patients with neurodegenerative disease to study excess mortality of the patients

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of neurodegenerative disease (ICD-10) in KUH or OUH between the years 2010-2021
* Age, sex and residency matched controls (Every research patient has 10 controls matched by age, gender, and place of residency)

Exclusion Criteria:

* Patients will be divided into different diagnostic groups based on the accepted diagnostic criteria in use. If some of the formed groups contain less than 5 subjects, the disease group in question is excluded from the analyses in order to ensure the privacy protection of the subjects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients admitted to Kuopio University Hospital (KUH) and Oulu University Hospital (OUH) Neurology outpatient clinic with a progressive neurodegenerative disease during 2010-2021 are identified from KUH and OUH data registry with all ICD-10 codes used in the diagnostics of neurodegenerative diseases. Their estimated number is 5572 patients. Clinical data of these patients are retrieved from the corresponding hospital data lakes. The patients will be divided into different diagnostic groups based on the accepted diagnostic criteria in use. Further, a matched control cohort is retrieved from the Finnish Population Information System maintained by the Digital and Population Data Services Agency. Every research patient has 10 controls matched by age, gender, and place of residency (according to the year of diagnosis), and the matching is performed for research patients that were alive at the end of the year of the diagnosis.
Sampling Method: Probability Sample
Enrollment: 61292 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Criminal behaviour: Type of offence, time of offence and other disruptive behaviour | 1996-2020
  Statistics Finland, Statistics on offences and coercive measures. Criminal behaviour is investigated utilising the reports of offences received by the police. The classification of offences is based on the three- or six-numbered offence classification by Statistics Finland, which enables the examination of different offences including e.g., violence, property, and traffic offences. The data extracted from the register include the type of the offence and time. Also, other disruptive behaviour based on the captures performed by the police (e.g., captures of intoxicated persons) is extracted.
Socio-demographic data | 1987-2021
  Employment, residency, Income, Marital status. Socio-demographic outcome data is extracted from Statistics Finland, FOLK Basic data module. Possible changes in employment and residency are examined, and mortality and emigration will be considered as censoring factors
Hospital diagnoses | 1994-2021
  Hospital diagnoses from the National Discharge Register. The National Discharge Register contains information of all hospitalizations after 1969, including ICD-8, ICD-9, and ICD-10 classifications to detect comorbidities of the patients. Two registers, "Terveydenhuollon hoitoilmoitusrekisteri (Hilmo)" and "Perusterveydenhuollon avohoidon hoitoilmoitus (Avohilmo)" of the Finnish Institute for Health and Welfare are used.
Medication use | 1995-2021
  Reimbursable drugs from the Social Insurance Institution of Finland (SII). Finnish residents are covered under the National Health Insurance (NHI) scheme run by the SII. SII maintains a nationwide registry of all patients, with dispensed reimbursable drugs 1995-, including opioids and neuropathic pain medications. Data of medication use, cost, and reimbursement data are gathered from the SII database.
Causes of death | 2010-2021
  Causes of death from Statistics Finland. Statistics Finland maintains a registry of causes of death and death certificates, which are supplemented with data from the population information system of the Population Register Centre. Registry data are used to study excess mortality of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No